CLINICAL TRIAL: NCT01793363
Title: Tracheostomy and Weaning From Mechanical Ventilation : Evaluation of the Lung Ultrasound Score
Acronym: TRAWELUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0144; 2012-A00366-37
Record Dates: First submitted 2013-02-07; First posted 2013-02-15 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Tracheotomy
Keywords: Tracheotomy; Weaning from mechanical ventilation; Lung ultrasound score
MeSH Terms: interventions — Tracheotomy

ARMS (1):
- tracheotomized patients (Experimental)
  Interventions: Procedure: Tracheotomy

INTERVENTIONS:
Procedure: Tracheotomy

SUMMARY:
Prospective, interventional multicentric study in ICU during weaning from mechanical ventilation in tracheotomized patients

DETAILED DESCRIPTION:
Prospective multicentric study on ICU evaluating Lung Ultrasound Score in tracheotomized patients during weaning from mechanical ventilation

ELIGIBILITY:
Inclusion Criteria:

* Adult patients tracheotomised during ICU stay
* Consent of patients

Exclusion Criteria:

* Tracheotomy before ICU
* No echogenicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Variation of lung ultrasound score | at day 1

SECONDARY OUTCOMES:
Time to weaning from mechanical ventilation | at day 1
Length of hospital stay | Day 1 + 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien PERBET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France